CLINICAL TRIAL: NCT04344288
Title: Corticosteroids During Covid-19 Viral Pneumonia Related to SARS-Cov-2 Infection
Acronym: CORTI-Covid
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Competent Authority's decision
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL20_0321; 2020-001553-48 (EudraCT Number)
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Viral Pneumonia Human Coronavirus; COVID-19
Keywords: Pneumology; viral pneumology; SARS-Cov-2; COVID 19; Prednisone
MeSH Terms: conditions — COVID-19 | interventions — Prednisone; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prednisone group (Experimental): Prednisone during 10 days after randomization
  Interventions: Drug: Prednisone
- Control group (Other)
  Interventions: Other: Control group

INTERVENTIONS:
Drug: Prednisone — The experimental group will receive oral prednisone during 10 days (0.75 mg/kg/day during 5 days then 20 mg/day during 5 more days)
  Arms: Prednisone group
Other: Control group — The control group will receive standard of care according to the international recommendations and practices of the investigational site. No corticosteroid therapy can be prescribed in this group.
  Arms: Control group

SUMMARY:
Infection with the SARS-Cov-2 virus, responsible of severe acute respiratory distress syndrome (SARS), is an emerging infectious disease called Covid-19 and declared as pandemic by the World Health Organization on March 11, 2020. This pandemic is responsible of significant mortality. In France, several thousand patients are hospitalized in intensive care units, and their number continues to increase. Mortality during Covid-19 is mainly linked to acute respiratory distress syndrome, which frequency is estimated in France to occur in 6% of infected patients. Comorbidities such as cardiovascular conditions, obesity and diabetes increase susceptibility to severe forms of Covid-19 and associated mortality. Therapeutic management has three components: symptomatic management, including supplementary oxygen therapy and in case of respiratory distress mechanical ventilation; the antiviral approach; and immunomodulation, aiming at reducing inflammation associated with viral infection, which is considered to take part in severe presentations of the disease.

During Covid-19 viral pneumonia related to SARS-COv-2, there is a significant release of pro-inflammatory cytokines in the acute phase of viral infection, which could participate in viral pneumonia lesions. In children with less mature immune system than adults, SARS-Cov-2 infection is less severe. The current prevailing assumption is that severe forms of Covid-19 may not only be related to high viral replication, but also to an excessive inflammatory response favoring acute lung injury and stimulating infection.

The investigators hypothesize that early control of the excessive inflammatory response may help reducing the risk of acute respiratory distress syndrome.

The investigators will evaluate the benefit, safety and tolerability of corticosteroid therapy to reduce the rate of subjects hospitalized for Covid-19 viral pneumonia who experience clinical worsening with a need of high-flow supplemental oxygen supplementation or transfer in intensive care units for respiratory support.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old,
* Hospitalization for COVID-19 infection confirmed by RT-PCR or other virological method,
* Peripheral saturation by pulse oximeter SpO2 ≤ 94% in ambient air measured twice at 5-15 min intervals, or PaO2 / FiO2 <300 mmHg,
* Abnormalities on the chest x-ray or CT scan suggestive of viral pneumonia,
* Signed informed consent by the patient.

Exclusion Criteria:

* Covid-19 infection with first symptoms lasting for more than 9 days according to the patient's interview; D1 of symptoms is defined by the first day with fever, cough, shortness of breath, and / or chills related to Covid-19 infection;
* Patients with primary or secondary immune deficiency, including: HIV, chronic hematological disease, solid organ transplant, ongoing immunosuppressive therapy,
* Long-term corticosteroid therapy defined by a prescription of more than 10 mg/d (prednisone equivalent),
* Suspected or confirmed infection with bacteria, fungal agents or viruses (in addition to Covid-19),
* Known contraindication to systemic corticosteroids,
* Systolic blood pressure <80 mmHg,
* SpO2 <90% under 5 L / min of oxygen using medium concentration mask, or higher oxygen requirements,
* Patient on long-term oxygen therapy,
* Ongoing mechanical ventilation,
* Ongoing septic shock ongoing,
* Ongoing multi-organ failure ongoing,
* Participating in other COVID-19 therapeutic clinical trial
* Pregnant or breast-feeding woman (oral diagnosis),
* No affiliation or beneficiary of health insurance,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-08-18 (Actual)

PRIMARY OUTCOMES:
Number of patients with a theoretical respiratory indication for transfer to intensive care unit evaluated by a SpO2 <90% stabilized at rest and under not more than 5 L / min of supplemental oxygen using medium concentration mask. | 7 days
  SpO2 <90% stabilized at rest and under not more than 5 L / min of supplemental oxygen using medium concentration mask. measured twice at 5-15 min intervalsThe average value of the two measurements will be calculated.

SECONDARY OUTCOMES:
disease severity assessed on a 7-level ordinal scale | 7 days
  level1: not hospitalized no limited activities, level 7: death
number of patients with a supplemental oxygen use | 7 days
radiological signs on chest imaging | 7 days
  Reduction of radiological signs on chest imaging
number of patients transferred to intensive care unit | 21 days
number of patients requiring invasive ventilation | 21 days
Duration of oxygen therapy | 21 days
  duration on days
number of adverse events induced by corticosteroid treatment | 21 days
number of patients with infections other than SARS-CoV-2 | 21 days
number of deaths | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François MORNEX, Principal Investigator — Hospices Civils de Lyon
Locations (12):
- France (12):
  - Hôpital Pneumologique et Cardiovasculaire Louis Pradel, Bron
  - CH Annecy-Genevois, Épagny
  - Groupement Hospitalier Nord, Lyon
  - Hôpital Edouard Herriot, Lyon
  - Hôpital St Joseph Saint Luc, Lyon
  - Hôpital St Joseph, Marseille
  - Centre hospitalier Lyon Sud, Pierre-Bénite
  - CHU St Etienne, Saint-Etienne
  - Clinique Charcot, Sainte-Foy-lès-Lyon
  - Clinique des Portes du Sud, Vénissieux
  - CHG Vienne, Vienne
  - Médipôle, Villeurbanne

IPD SHARING:
Plan to Share IPD: Undecided